CLINICAL TRIAL: NCT02702661
Title: Fascia Iliaca Compartment Block and Local Anaesthetic Infiltration for Pain Control Following Hip Arthroscopic Surgery
Brief Title: PRCT of FICB vs LAI for Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Vikas Khanduja MA FRCS (Orth), Consultant Orthopaedic Surgeon & Associate Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A092336
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Femoroacetabular Impingement
Keywords: Fascia Iliaca Block; Local Anaesthetic Infiltration; Hip Arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Procedure - FICB (Experimental): Fascia Iliaca Block following Hip Arthroscopy - Drug - Levobupivacaine 0.125% - 40ml
  Interventions: Procedure: Fascia Iliaca Compartment Block (FICB); Drug: Levobupivacaine
- Procedure - LAI (Active Comparator): Local Anaesthetic Infiltration following Hip Arthroscopy - Drug - Levobupivacaine 0.125% - 40ml
  Interventions: Procedure: Local Anaesthetic Infiltration (LAI); Drug: Levobupivacaine

INTERVENTIONS:
Procedure: Fascia Iliaca Compartment Block (FICB) — Fascia Iliaca Compartment Block
  Arms: Procedure - FICB
Procedure: Local Anaesthetic Infiltration (LAI) — Local Anaesthetic Infiltration (LAI) of the portal tracts
  Arms: Procedure - LAI
Drug: Levobupivacaine — Levobupivacaine 0.125% - 40ml

SUMMARY:
A prospective randomised controlled trial involving patients undergoing hip arthroscopy. Participants were randomised to receiving either Fascia Iliaca Compartment Block (FICB) or Local Anaesthetic Infiltration (LAI) of the portal tracts with local anaesthetic. Supplemental analgesia was also used in both groups on an on-demand basis. Pain level is assessed at 1,3,6, and 24 hours post surgery. The primary outcome measure was the post-operative level of pain as assessed by Numeric Pain Score 6 hours after surgery. Secondary outcome measures were the frequency and the dose of morphine and other medications consumed at 1 and 24 hours after surgery as well as any other adverse events relating to pain or medications used for pain relief in both the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years
* Primary elective hip arthroscopy on a native hip for combined soft tissue injuries and FAI pathology
* Able to read, write and communicate in English

Exclusion Criteria:

* Patients who did not want to be involved in the Trial
* Unable to give informed consent
* Previous hip surgery
* Patients younger than 18 years of age
* Chronic opioids users
* Patients known to have an allergy or intolerance to local anaesthetic agents or none steroidal anti-inflammatory medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Level of pain as assessed by Numeric Pain Score | 6 hours after surgery

SECONDARY OUTCOMES:
Frequency of morphine consumed | 1 and 24 hours after surgery
Total dose of morphine consumed | 1 and 24 hours after surgery
Total dose of codeine consumed | 1 and 24 hours after surgery
Nausea and Vomiting | 1 and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Khanduja, MA, FRCS (Orth), Study Director — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No